CLINICAL TRIAL: NCT02983708
Title: Neuroregenerative Potential of Intravenous G-CSF and Autologous Peripheral Blood Stem Cells in Children With Cerebral Palsy: a Randomized, Double-blind Cross-over Study
Brief Title: Neuroregenerative Potential of Intravenous G-CSF and Autologous Peripheral Blood Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Ho Lee, Professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-PB-2011
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Neurodegeneration; G-CSF; Peripheral Blood Mononuclear Cells; Cerebral Palsy
Keywords: Neuroregeneration; G-CSF; Peripheral blood mononuclear cells; Cerebral palsy
MeSH Terms: conditions — Nerve Degeneration; Cerebral Palsy | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mPBMC group (Experimental): G-CSF would be administered for 5 days and then mobilized peripheral blood mononuclear cells (mPBMCs) would be collected in all included patients. One month after cryopreservation of the mPBMCs (M1), patients will be randomized to receive either mPBMCs or placebo. Six months after randomization (M7), cross-over infusion of mPBMCs or placebo will be performed and the patients are observed for another 6 months. mPBMCs group would be included all patients who received mPBMCs at M1 or M7.
  Interventions: Biological: Peripheral blood mononuclear cells (mPBMC); Drug: G-CSF
- Placebo group (Placebo Comparator): G-CSF would be administered for 5 days and then mobilized peripheral blood mononuclear cells (mPBMCs) would be collected in all included patients. One month after cryopreservation of the mPBMCs (M1), patients will be randomized to receive either mPBMCs or placebo. Six months after randomization (M7), cross-over infusion of mPBMCs or placebo will be performed and the patients are observed for another 6 months. Placebo group would be included all patients who received placebo at M1 or M7.
  Interventions: Drug: G-CSF; Drug: Placebo

INTERVENTIONS:
Biological: Peripheral blood mononuclear cells (mPBMC)
  Arms: mPBMC group
Drug: G-CSF
Drug: Placebo
  Arms: Placebo group

SUMMARY:
The current study describes a randomized, double-blind, cross-over study of intravenous G-CSF followed by infusion with autologous mobilized peripheral blood mononuclear cells (mPBMCs) in children with cerebral palsy (CP) to determine the safety and feasibility of the procedure, as well as the potential efficacy for improving neurological impairment.

DETAILED DESCRIPTION:
We hypothesized that mobilized peripheral blood mononuclear cells (mPBMCs) would be a better source of cell therapy for children with CP, if these cells had a similar neuroregenerative potential to bone marrow/cord blood mononuclear cells (MNCs). Multipotent precursor cells exist in peripheral blood, and a fraction of elutriated blood cells from normal individuals contains MNCs that have the potential to be MSCs. There are several advantages to using mPBMCs for cell therapy in children with CP: the G-CSF that is used to mPBMCs has neuroregenerative potential; the collection and fractionation of stem cells can be repeated; and, the therapy is suitable for most children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Non severe type of cerebral palsy
* Evidences of abnormal MRI findings such as periventricular leukomalacia
* Collected mobilized peripheral blood mononuclear cell counts > 1×10^8/kg or CD34+ cell counts > 1×10^6/kg
* Consent form

Exclusion Criteria:

* Previous trials of autologous cord blood infusion or erythropoietin/G-CSF
* Chromosomal abnormalities

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Overall improvement as a score changes in GMFM > 4 points | 6 months

IPD SHARING:
Plan to Share IPD: Undecided
We have to get individual permissions to make IPD available to other researchers.

REFERENCES:
- [Derived] Rah WJ, Lee YH, Moon JH, Jun HJ, Kang HR, Koh H, Eom HJ, Lee JY, Lee YJ, Kim JY, Choi YY, Park K, Kim MJ, Kim SH. Neuroregenerative potential of intravenous G-CSF and autologous peripheral blood stem cells in children with cerebral palsy: a randomized, double-blind, cross-over study. J Transl Med. 2017 Jan 21;15(1):16. doi: 10.1186/s12967-017-1120-0. PMID 28109298